CLINICAL TRIAL: NCT01569971
Title: Adolescent, Caregiver, and Young Adult Perspectives of the Transition From Pediatric to Adult Care for Sickle Cell Disease: A Preliminary Evaluation of the Sickle Cell Disease Transition Program
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Plough Foundation (Unknown); Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: XPD12-025 TRANSCD; U1EMC19331 (Other Grant/Funding Number: Health Resources and Services Administration)
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Sickle Cell Disease
Keywords: Transition Program; Perspectives
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Restraint, Physical; Focus Groups; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Adolescents: Adolescents with SCD (all genotypes) age 12 years old up to 18 years old and currently receiving services through the St. Jude Children's Research Hospital Sickle Cell Disease Transition Program.
  Interventions: Other: Assessment
- Caregivers: Caregiver of an adolescent with SCD who has resided with the adolescent for at least two years prior.
  Interventions: Other: Assessment
- Young Adults: Young adults with SCD (all genotypes) age equal to 18 years up to and equal to 30 years of age who have transitioned to adult care.
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — In this study, through the use of focus groups and questionnaires, we will identify perceptions of transition from pediatric to adult care, transition readiness, disease knowledge, and self-management skills, and assess components of the St. Jude Children's Research Hospital (SJCRH) Sickle Cell Disease Transition Program. Participants will participate in focus groups to discuss transition and transition-related concepts and evaluate components of the transition program. Additionally, participants will complete questionnaires about specific aspects of the transition program and about current disease knowledge and management skills.
  Other Names: Focus Groups; Questionnaires

SUMMARY:
Sickle cell disease (SCD) is a debilitating genetic disorder affecting 70,000-100,000 Americans. It is frequently associated with very serious medical complications. For children with SCD, successfully transitioning to adult care is a vital step in ensuring continuity of care, managing their disease, and improving their health outcomes. Transition programs have been created to facilitate the transition process. However, few studies have assessed transition readiness and whether transition program components meet the transition needs of patients and families.

The purpose of this study is to explore transitioning from pediatric care to adult care and to assess components of the SJCRH SCD Transition Program from three perspectives: adolescents with SCD, their caregivers, and young adults with SCD who have transitioned to adult care. Data collection methods will include focus groups, questionnaires, and checklists. Qualitative data analysis procedures will be used to examine the data.

DETAILED DESCRIPTION:
In this study, through the use of focus groups and questionnaires, we will identify perceptions of transition from pediatric to adult care, transition readiness, disease knowledge, and self-management skills, and assess components of the St. Jude Children's Research Hospital (SJCRH) Sickle Cell Disease Transition Program. Participants will participate in focus groups to discuss transition and transition-related concepts and evaluate components of the transition program. Additionally, participants will complete questionnaires about specific aspects of the transition program and about current disease knowledge and management skills.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with SCD (all genotypes) ages ≥ 12 years old and ≤ 18 years old and currently receiving services through the SJCRH Sickle Cell Disease Transition Program.
* Caregivers who have resided with the adolescent with SCD for at least 2 years prior.
* Young adults with SCD (all genotypes) ages ≥ 18 years old and ≤ 30 years old who have transitioned to adult care

Exclusion Criteria:

* Non-English speakers.
* Adolescents and young adults with sickle cell trait.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 1. Adolescents with SCD (all genotypes) ages ≥ 12 years old and ≤ 18 years old and currently receiving services through the SJCRH Sickle Cell Disease Transition Program
  2. Caregiver of an adolescent with SCD who has resided with the adolescent for at least 2 years prior
  3. Young adults with SCD (all genotypes) ages ≥ 18 years old and ≤ 30 years old who have transitioned to adult care
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Grounded theory qualitative analysis of data | 1 day
  First, data will be prepared for qualitative analysis. Digital audio files from the focus groups will be transcribed verbatim and questionnaire data will be entered into an Excel data file. Second, focus group data will be qualitatively analyzed using the constant comparative process. A qualitative data analysis program, NVivo9 (Victoria, Australia) will be used to assist with this coding process.

CONTACTS AND LOCATIONS:
Overall Officials: Jerlym Porter, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols